CLINICAL TRIAL: NCT02698982
Title: Impact of Tight Intraoperative Blood Pressure and Depth of Anesthesia Control on the Incidence of Postoperative Cognitive Impairment in Elderly Patients
Brief Title: Optimized Anesthesia to Reduce Postoperative Cognitive Impairment in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Céline Boudart, MD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P2015/539
Record Dates: First submitted 2016-02-12; First posted 2016-03-04 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Elderly ; Moderate Risk Surgery
Keywords: elderly; postoperative cognitive dysfunction; postoperative delirium; depth of anesthesia; intraoperative blood pressure monitoring
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Monitoring (Experimental): Elderly scheduled for moderate risk surgery Depth of anesthesia monitoring and Continuous non invasive blood pressure monitoring accessible to the anesthesia provider.
  Interventions: Device: Depth of anesthesia monitoring (BIS, Covidien USA) and Continus non invasive blood pressure monitoring (Clearsight, Edwards LifeScience, USA); Procedure: moderate risk surgery
- Sham (Sham Comparator): Elderly scheduled for moderate risk surgery Depth of anesthesia monitoring and Continuous non invasive blood pressure monitoring blinded to the anesthesia provider
  Interventions: Procedure: moderate risk surgery
- Control (No Intervention): elderly non scheduled for surgery

INTERVENTIONS:
Device: Depth of anesthesia monitoring (BIS, Covidien USA) and Continus non invasive blood pressure monitoring (Clearsight, Edwards LifeScience, USA)
  Arms: Monitoring
Procedure: moderate risk surgery
  Arms: Monitoring; Sham

SUMMARY:
The aim of this study is to demonstrate that in elderly and frail patients, a narrower control of intraoperative blood pressure (BP) by the use of a continuous and noninvasive BP monitoring, coupled with an adequate depth of anesthesia, will reduce the incidence of postoperative cognitive impairment and the hospital length of stay.

DETAILED DESCRIPTION:
Postoperative cognitive impairment (delirium and cognitive dysfunction) are frequent and feared complications in the elderly; they increase the postoperative morbidity and mortality, worsen the cognitive and functional outcome with loss of independence and increase the hospitalization length and costs . However, the etiology of these postoperative cognitive impairment, although probably multifactorial, remains unclear and strongly debated.

The investigators hypothesize that excessive anesthesia depths associated with intraoperative hypotension may play a critical role in the pathogenesis of cognitive impairment following surgery.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (over the age of 70) undergoing elective moderate risk surgery requiring a general anesthesia
* Patients who provide written informed consent
* patient fluent in french

Exclusion Criteria:

* Patients under 70 years of age
* Surgery under locoregional anesthesia or emergent surgery or minor risk surgery
* Patients requiring invasive blood pressure monitoring (for medical reason or high risk surgery)
* Patients with arrhythmia and/or atrial fibrillation
* Patients with preoperative delirium or cognitive dysfunction (moca test < 26)
* Patients not fluent in French
* Patients without the capacity to give written informed consent or refusal of consent
* Patients undergoing surgery or included in another protocol within 3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
postoperative delirium detected by the Confusion Assessment Method (CAM) | 3 day postoperative
  Screening of postoperative delirium by the CAM, every day until the 3rd postoperative day

SECONDARY OUTCOMES:
postoperative change in cognitive function detected by a battery of neuropsychological test. | baseline and 1 week and 3 month postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Obbergh, MD PhD, Study Director — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium